CLINICAL TRIAL: NCT03961009
Title: A Phase III, Open-label, Prospective, Multicenter Study to Assess Efficacy, Safety and Pharmacokinetics of Kedrion Intravenous Immunoglobulin (IVIg) 10% in Primary Immunodeficiency Disease (PID) Patients
Brief Title: Clinical Assessment of Pharmacokinetics, Efficacy, and Safety of 10% IVIg in PID Patients
Acronym: CARES10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kedrion S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIG10_US3_PID01
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Primary Immunodeficiency Disease
Keywords: Immunoglobulin; Kedrion IVIg10%; IgG antibodies; Agammaglobulinemia; Hypogammaglobulinemia
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Agammaglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Kedrion IVIG 10% (Experimental): Participants received intravenous infusion of Kedrion IVIG 10% at a dose of 200 to 800 milligrams per kilogram (mg/kg) body weight on every 21 or 28 days for period of 48 weeks.
  Interventions: Biological: Kedrion IVIG 10%

INTERVENTIONS:
Biological: Kedrion IVIG 10% — Kedrion intravenous immunoglobulin (IVIg) 10%

SUMMARY:
The purpose of this study was to assess efficacy and safety of Kedrion Immunoglobulin 10% (KIg10) in participants with Primary Immunodeficiency (PID).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent obtained from participant/participant's parent(s) or legally acceptable representative indicating that they understand the purpose of and procedures required for the study and are willing to participate in it.
* Confirmed clinical diagnosis of a PID, requiring treatment with IVIg and have documented agammaglobulinemia (defined as the total absence of one or more classes of antibodies) or hypogammaglobulinemia (defined as low levels of one or more classes [that is at least 2 standard deviations under the mean level per age])
* Male or female, ages 2 to 70 years at screening
* Received 200 to 800 mg/kg of a commercially available IVIg therapy in the range of 21- or 28-day intervals (±3 days or ±4 days, respectively) for at least 3 infusion cycles prior to screening
* At least 2 documented IgG trough levels while receiving an IVIg, of greater than or equals to (>=) 6 gram per liter (g/L) obtained at 2 infusion cycles within 12 months (1 must be within 6 months) prior to Informed Consent Form (ICF) signature
* Participant is willing to comply all requirements of the protocol.
* Females of child-bearing potential with a negative urine pregnancy test and who agree to employ adequate birth control measures during the study
* Authorization to access personal health information
* Participant previously participating in a clinical trial with another experimental IVIg may be enrolled if they have received stable commercially available IVIg therapy for at least 3 infusion cycles (21 or 28 days) prior to screening
* Participant currently on treatment with any subcutaneous immunoglobulin (SCIG) can be enrolled if they are switched to stable commercially available IVIg therapy for at least 3 infusion cycles (21 or 28 days) prior to screening

Exclusion Criteria:

* Newly diagnosed PID and and naïve to IgG replacement therapy
* Dysgammaglobulinemia (defined as a deficiency in one or more classes of antibodies, but not severe enough to require substitutive therapy) or isolated IgG subclass deficiency or profound primary T-cell deficiency (defined as the absence or severe reduction of T lymphocytes [CD3+ <300 cells per cubic millimeter (cell/mm3)] and an absent or particularly low proliferative response [10% of the lower normal range] to phytohaemagglutinin P [PHA])
* Has history of severe or serious reactions or hypersensitivity to IVIg or other injectable forms of IgG
* Has history of thrombotic events (including deep vein thrombosis, cerebrovascular accident, pulmonary embolism, transient ischemic attacks, or myocardial infarction), as defined by at least 1 event in participant's lifetime
* Has IgA deficiency with documented antibodies to IgA
* Have received blood products that have not undergone viral inactivation measures within 12 months prior to Informed Consent Form (ICF) signature
* Has significant protein losing enteropathy, nephrotic syndrome, or lymphangiectasia
* Has an acute infection as documented by culture or diagnostic imaging and/or a body temperature >= 38 degree Celsius (°C) (>=100.4 degree Fahrenheit (°F) within 7 days prior to screening
* Has acquired immunodeficiency syndrome (AIDS) and/or hepatitis B/C active disease at ICF signature
* Has levels of Alanine aminotransferase (ALT) or aspartate aminotransferase (AST), 2.5 times of the upper limit of normal for the laboratory designated for the study
* Using an implanted venous access device
* Has profound anemia (haemoglobin less than10 gram per deciliter [g/dl]) or persistent severe neutropenia (<= 1000 neutrophils per millimeter cube (mm^3) or lymphopenia of less than 500 cells per microliter
* Have severe chronic condition such as renal failure (creatinine concentration > 2.0 times the upper limit of normal) with proteinuria, congestive heart failure (New York Heart Association III/IV), cardiomyopathy, cardiac arrhythmia associated with thromboembolic events (e.g., atrial fibrillation), unstable or advanced ischemic heart disease, hyper viscosity, or any other condition that the Investigator believes is likely to interfere with evaluation of the study drug or with satisfactory conduct of the trial. Normal values for serum creatinine are the following: a) Female (18+ years): 45 - 84 micromole per liter (mcmol/L) or 0.51 - 0.95 milligrams per deciliter (mg/dl); b) Male (18+ years): 59 - 103 mcmol/L or 0.67 - 1.17 mg/dl
* Has history of a malignant disease other than properly treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin within 24 months prior to ICF signature
* Has history of pharmacoresistant epilepsy or multiple episodes of migraine (defined as at least 1 episode within 6 months of ICF signature) not completely controlled by medication
* Participants must not be receiving steroids (oral or parenteral daily dose of >= 0.15 milligram per kilogram per day (mg/kg/day) of prednisone or equivalent) or other immunosuppressive drugs or chemotherapy
* Females who are pregnant, breast feeding or planning a pregnancy during the course of the study. Women who become pregnant during the study will be withdrawn from the study
* Has participated in another clinical study within 3 weeks prior to study ICF signature
* Has history of drug or alcohol abuse within the 6 months before screening
* Has Employed or a direct relative of an employee of the CRO, the study site, or the Sponsor
* Previously treated under this protocol
* Unable to provide informed consent or provide informed consent by a legally authorized representative

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Kedrion SpA
Locations (11):
- United States (11):
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Dr. Henry J. Kanarek - Allergy, Asthma & Immunology, Overland Park, Kansas
  - Midwest Immunology Clinic and Infusion Center, Plymouth, Minnesota
  - Allergy and Immunology Associates, Little Silver, New Jersey
  - University of Buffalo, Buffalo, New York
  - Optimed Research, Columbus, Ohio
  - Ohio Clinical Research Associates, Inc., Mayfield Heights, Ohio
  - Toledo Institute of Clinical Research Inc, Toledo, Ohio
  - Allergy Partners of North Texas Research, Dallas, Texas
  - AARA Research Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 11 sites in the United States from 30 April 2019 (first participant first visit) to 21 December 2020 (last participant last visit).
Pre-assignment Details: A total of 59 participants were screened, out of which 47 participants were enrolled and received the treatment in this study.
Period: Overall Study
Arm/Group | Kedrion IVIG 10%
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who had received at least 1 dose of study medication.
Groups:
- Kedrion IVIG 10%: Participants received intravenous infusion of Kedrion IVIG 10% at a dose of 200 to 800 mg/kg body weight on every 21 or 28 days for period of 48 weeks.
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45
  Mexican | 1
  White and African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Acute Serious Bacterial Infections (ABSIs)
Description: Incidence rate was defined as the mean number of acute serious bacterial infections (bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, visceral abscess, osteomyelitis/septic arthritis) per participant-year according to pre-specified criteria.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: The FAS included all participants who had received at least 1 dose of study medication. Here, "Number Analyzed" signifies those participants who were evaluable at specified time points as per the dosing schedule.
Measure: Mean (Standard Deviation); unit: infections per participant-year
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
infections per participant-year
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 0.0 (0.0)
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 0.0 (0.0)

2. Secondary Outcome: Serum Immunoglobulin G (IgG) Trough Levels
Description: The serum IgG trough levels were collected and analyzed at a central laboratory.
Time Frame: At baseline, Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who have received at least 1 dose of study medication. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per the dosing schedule.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
grams per liter (g/L)
  Baseline | 10.317 (3.1342)
  21-day dosing schedule: Week 51: number analyzed (Participants) | 8
  21-day dosing schedule: Week 51 | 11.433 (1.7935)
  28-day dosing schedule: Week 52: number analyzed (Participants) | 39
  28-day dosing schedule: Week 52 | 10.297 (2.1167)

3. Secondary Outcome: Immunoglobulin G (IgG) Subclasses Levels (IgG1, IgG2, IgG3, IgG4)
Description: IgG subclasses levels (IgG1, IgG2, IgG3, IgG4) were collected and analyzed at a central laboratory.
Time Frame: At baseline, Weeks 16, 32 and 48 (28-day dosing schedule); Weeks 18, 30, 48 (21-day dosing schedule)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
g/L
  IgG1: Baseline | 5.798 (1.7504)
  IgG1: 28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  IgG1: 28-day dosing schedule: Week 16 | 5.605 (1.6115)
  IgG1: 21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  IgG1: 21-day dosing schedule: Week 18 | 5.968 (1.5094)
  IgG1: 28-day dosing schedule: Week 32: number analyzed (Participants) | 39
  IgG1: 28-day dosing schedule: Week 32 | 5.679 (1.3965)
  IgG1: 21-day dosing schedule: Week 30: number analyzed (Participants) | 8
  IgG1: 21-day dosing schedule: Week 30 | 5.979 (0.9430)
  IgG1: 28-day dosing schedule: Week 48: number analyzed (Participants) | 37
  IgG1: 28-day dosing schedule: Week 48 | 5.634 (1.4139)
  IgG1: 21-day dosing schedule: Week 48: number analyzed (Participants) | 8
  IgG1: 21-day dosing schedule: Week 48 | 6.210 (0.9430)
  IgG2: Baseline | 3.527 (0.9635)
  IgG2: 28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  IgG2: 28-day dosing schedule: Week 16 | 3.419 (0.8803)
  IgG2: 21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  IgG2: 21-day dosing schedule: Week 18 | 4.113 (1.0155)
  IgG2: 28-day dosing schedule: Week 32: number analyzed (Participants) | 39
  IgG2: 28-day dosing schedule: Week 32 | 3.458 (0.7705)
  IgG2: 21-day dosing schedule: Week 30: number analyzed (Participants) | 8
  IgG2: 21-day dosing schedule: Week 30 | 4.079 (0.4975)
  IgG2: 28-day dosing schedule: Week 48: number analyzed (Participants) | 37
  IgG2: 28-day dosing schedule: Week 48 | 3.475 (0.7848)
  IgG2: 21-day dosing schedule: Week 48: number analyzed (Participants) | 8
  IgG2: 21-day dosing schedule: Week 48 | 4.234 (0.5649)
  IgG3: Baseline | 0.405 (0.3109)
  IgG3: 28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  IgG3: 28-day dosing schedule: Week 16 | 0.351 (0.3459)
  IgG3: 21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  IgG3: 21-day dosing schedule: Week 18 | 0.271 (0.1239)
  IgG3: 28-day dosing schedule: Week 32: number analyzed (Participants) | 39
  IgG3: 28-day dosing schedule: Week 32 | 0.352 (0.3461)
  IgG3: 21-day dosing schedule: Week 30: number analyzed (Participants) | 8
  IgG3: 21-day dosing schedule: Week 30 | 0.249 (0.0885)
  IgG3: 28-day dosing schedule: Week 48: number analyzed (Participants) | 37
  IgG3: 28-day dosing schedule: Week 48 | 0.329 (0.3268)
  IgG3: 21-day dosing schedule: Week 48: number analyzed (Participants) | 8
  IgG3: 21-day dosing schedule: Week 48 | 0.253 (0.0658)
  IgG4: Baseline | 0.2213 (0.12779)
  IgG4: 28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  IgG4: 28-day dosing schedule: Week 16 | 0.2388 (0.09656)
  IgG4: 21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  IgG4: 21-day dosing schedule: Week 18 | 0.2744 (0.06415)
  IgG4: 28-day dosing schedule: Week 32: number analyzed (Participants) | 39
  IgG4: 28-day dosing schedule: Week 32 | 0.2425 (0.09290)
  IgG4: 21-day dosing schedule: Week 30: number analyzed (Participants) | 8
  IgG4: 21-day dosing schedule: Week 30 | 0.2838 (0.06412)
  IgG4: 28-day dosing schedule: Week 48: number analyzed (Participants) | 37
  IgG4: 28-day dosing schedule: Week 48 | 0.2396 (0.09355)
  IgG4: 21-day dosing schedule: Week 48: number analyzed (Participants) | 8
  IgG4: 21-day dosing schedule: Week 48 | 0.2950 (0.05381)

4. Secondary Outcome: Number of Participants With Total Immunoglobulin G (IgG) Trough Levels Less Than or Equal to (<=) 6 Grams/Liter (g/L) Criteria
Description: Number of participants with Total IgG trough levels <= 6 g/L criteria were reported.
Time Frame: Up to 12 months
Population: FAS included all participants who have received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants | 1

5. Secondary Outcome: Anti-Tetanus Toxoid Antibody Levels
Description: The anti-tetanus toxoid antibody levels were collected and analyzed at a central laboratory. This antibody level was measured in international units per milliliter (IU/mL).
Time Frame: Baseline, Weeks 16, 32 and 48 (28-day dosing schedule); Weeks 18, 30, 48 (21-day dosing schedule)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
IU/mL
  Baseline | 2.526 (1.4158)
  28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16 | 2.589 (2.0770)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18 | 2.654 (0.9853)
  28-day dosing schedule: Week 32: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32 | 2.345 (0.8820)
  21-day dosing schedule: Week 30: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30 | 2.643 (0.9374)
  28-day dosing schedule: Week 48: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48 | 2.207 (0.8565)
  21-day dosing schedule: Week 48: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48 | 3.299 (1.3307)

6. Secondary Outcome: Anti-Pneumococcal Capsular Polysaccharide Antibody Levels
Description: Anti-pneumococcal capsular polysaccharide antibody levels for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 were collected and analyzed at a central laboratory.
Time Frame: Baseline, Weeks 16, 32 and 48 (28-day dosing schedule); Weeks 18, 30, 48 (21-day dosing schedule)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
milligrams per liter (mg/L)
  Baseline: Serotype 1 | 2.66 (4.820)
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 1 | 1.55 (1.481)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 1 | 4.89 (5.740)
  28-day dosing schedule: Week 32: Serotype 1: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 1 | 1.66 (2.114)
  21-day dosing schedule: Week 30: Serotype 1: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 1 | 4.74 (5.692)
  28-day dosing schedule: Week 48: Serotype 1: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 1 | 1.49 (1.707)
  21-day dosing schedule: Week 48: Serotype 1: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 1 | 4.28 (4.926)
  Baseline: Serotype 12: number analyzed (Participants) | 43
  Baseline: Serotype 12 | 0.81 (1.103)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 35
  28-day dosing schedule: Week 16: Serotype 12 | 0.75 (1.201)
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 12 | 0.58 (0.175)
  28-day dosing schedule: Week 32: Serotype 12: number analyzed (Participants) | 29
  28-day dosing schedule: Week 32: Serotype 12 | 0.86 (1.280)
  21-day dosing schedule: Week 30: Serotype 12: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 12 | 0.55 (0.120)
  28-day dosing schedule: Week 48: Serotype 12: number analyzed (Participants) | 27
  28-day dosing schedule: Week 48: Serotype 12 | 0.82 (1.159)
  21-day dosing schedule: Week 48: Serotype 12: number analyzed (Participants) | 7
  21-day dosing schedule: Week 48: Serotype 12 | 0.59 (0.090)
  Baseline: Serotype 14 | 9.04 (20.383)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 14 | 11.88 (29.791)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 14 | 6.11 (3.302)
  28-day dosing schedule: Week 32: Serotype 14: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 14 | 11.96 (26.509)
  21-day dosing schedule: Week 30: Serotype 14: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 14 | 5.76 (2.752)
  28-day dosing schedule: Week 48: Serotype 14: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 14 | 13.02 (34.794)
  21-day dosing schedule: Week 48: Serotype 14: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 14 | 6.14 (3.408)
  Baseline: Serotype 17 | 2.55 (4.249)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 17 | 2.08 (3.977)
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 17 | 3.25 (3.146)
  28-day dosing schedule: Week 32: Serotype 17: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 17 | 1.89 (2.952)
  21-day dosing schedule: Week 30: Serotype 17: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 17 | 3.38 (4.058)
  28-day dosing schedule: Week 48: Serotype 17: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 17 | 1.76 (3.043)
  21-day dosing schedule: Week 48: Serotype 17: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 17 | 3.09 (3.111)
  Baseline: Serotype 19 | 3.71 (5.275)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 19 | 4.95 (8.597)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 19 | 3.20 (1.074)
  28-day dosing schedule: Week 32: Serotype 19: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 19 | 3.71 (4.200)
  21-day dosing schedule: Week 30: Serotype 19: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 19 | 2.88 (0.686)
  28-day dosing schedule: Week 48: Serotype 19: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 19 | 4.25 (7.328)
  21-day dosing schedule: Week 48: Serotype 19: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 19 | 2.86 (0.958)
  Baseline: Serotype 2 | 2.38 (2.294)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 2 | 2.04 (1.618)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 2 | 3.34 (3.701)
  28-day dosing schedule: Week 32: Serotype 2: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 2 | 2.11 (1.502)
  21-day dosing schedule: Week 30: Serotype 2: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 2 | 3.48 (4.071)
  28-day dosing schedule: Week 48: Serotype 2: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 2 | 2.01 (1.283)
  21-day dosing schedule: Week 48: Serotype 2: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 2 | 3.35 (3.342)
  Baseline: Serotype 20 | 2.71 (2.296)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 20 | 2.63 (3.007)
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 20 | 3.05 (1.425)
  28-day dosing schedule: Week 32: Serotype 20: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 20 | 2.76 (3.153)
  21-day dosing schedule: Week 30: Serotype 20: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 20 | 3.16 (1.614)
  28-day dosing schedule: Week 48: Serotype 20: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 20 | 2.51 (2.779)
  21-day dosing schedule: Week 48: Serotype 20: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 20 | 3.05 (1.295)
  Baseline: Serotype 22 | 1.33 (1.968)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 22 | 0.84 (0.938)
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 22 | 2.36 (3.554)
  28-day dosing schedule: Week 32: Serotype 22: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 22 | 0.83 (0.698)
  21-day dosing schedule: Week 30: Serotype 22: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 22 | 2.78 (4.627)
  28-day dosing schedule: Week 48: Serotype 22: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 22 | 0.88 (0.670)
  21-day dosing schedule: Week 48: Serotype 22: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 22 | 2.51 (3.652)
  Baseline: Serotype 23 | 1.65 (2.336)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 38
  28-day dosing schedule: Week 16: Serotype 23 | 1.42 (2.501)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 23 | 1.28 (0.696)
  28-day dosing schedule: Week 32: Serotype 23: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 23 | 1.37 (2.064)
  21-day dosing schedule: Week 30: Serotype 23: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 23 | 1.34 (0.607)
  28-day dosing schedule: Week 48: Serotype 23: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 23 | 1.47 (2.270)
  21-day dosing schedule: Week 48: Serotype 23: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 23 | 1.50 (0.733)
  Baseline: Serotype 26 | 1.72 (1.910)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 38
  28-day dosing schedule: Week 16: Serotype 26 | 1.32 (1.578)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 26 | 1.83 (2.050)
  28-day dosing schedule: Week 32: Serotype 26: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 26 | 1.36 (1.515)
  21-day dosing schedule: Week 30: Serotype 26: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 26 | 1.70 (1.505)
  28-day dosing schedule: Week 48: Serotype 26: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 26 | 1.39 (1.549)
  21-day dosing schedule: Week 48: Serotype 26: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 26 | 1.73 (1.482)
  Baseline: Serotype 3 | 2.41 (5.964)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 3 | 1.41 (2.362)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 3 | 4.74 (7.812)
  28-day dosing schedule: Week 32: Serotype 3: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 3 | 1.42 (2.526)
  21-day dosing schedule: Week 30: Serotype 3: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 3 | 4.24 (6.480)
  28-day dosing schedule: Week 48: Serotype 3: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 3 | 1.12 (1.287)
  21-day dosing schedule: Week 48: Serotype 3: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 3 | 4.69 (7.854)
  Baseline: Serotype 34 | 1.83 (2.663)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 34 | 1.34 (1.718)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 34 | 3.33 (4.843)
  28-day dosing schedule: Week 32: Serotype 34: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 34 | 1.30 (1.524)
  21-day dosing schedule: Week 30: Serotype 34: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 34 | 3.73 (6.610)
  28-day dosing schedule: Week 48: Serotype 34: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 34 | 1.35 (1.585)
  21-day dosing schedule: Week 48: Serotype 34: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 34 | 3.04 (4.276)
  Baseline: Serotype 4: number analyzed (Participants) | 32
  Baseline: Serotype 4 | 0.88 (1.366)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 25
  28-day dosing schedule: Week 16: Serotype 4 | 0.54 (0.896)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 7
  21-day dosing schedule: Week 18: Serotype 4 | 0.57 (0.576)
  28-day dosing schedule: Week 32: Serotype 4: number analyzed (Participants) | 10
  28-day dosing schedule: Week 32: Serotype 4 | 1.07 (1.292)
  21-day dosing schedule: Week 30: Serotype 4: number analyzed (Participants) | 5
  21-day dosing schedule: Week 30: Serotype 4 | 0.66 (0.434)
  28-day dosing schedule: Week 48: Serotype 4: number analyzed (Participants) | 12
  28-day dosing schedule: Week 48: Serotype 4 | 0.89 (1.187)
  21-day dosing schedule: Week 48: Serotype 4: number analyzed (Participants) | 5
  21-day dosing schedule: Week 48: Serotype 4 | 0.68 (0.466)
  Baseline: Serotype 43 | 1.36 (0.713)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 43 | 1.07 (0.665)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 43 | 1.51 (0.645)
  28-day dosing schedule: Week 32: Serotype 43: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 43 | 1.08 (0.568)
  21-day dosing schedule: Week 30: Serotype 43: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 43 | 1.43 (0.468)
  28-day dosing schedule: Week 48: Serotype 43: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 43 | 1.12 (0.605)
  21-day dosing schedule: Week 48: Serotype 43: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 43 | 1.61 (0.482)
  Baseline: Serotype 5 | 3.64 (5.551)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 5 | 2.68 (3.650)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 5 | 6.56 (9.390)
  28-day dosing schedule: Week 32: Serotype 5: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 5 | 2.65 (3.081)
  21-day dosing schedule: Week 30: Serotype 5: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 5 | 6.51 (10.172)
  28-day dosing schedule: Week 48: Serotype 5: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 5 | 2.44 (3.145)
  21-day dosing schedule: Week 48: Serotype 5: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 5 | 5.41 (7.414)
  Baseline: Serotype 51 | 2.82 (5.468)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 51 | 1.66 (0.777)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 51 | 5.96 (8.691)
  28-day dosing schedule: Week 32: Serotype 51: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 51 | 1.65 (0.786)
  21-day dosing schedule: Week 30: Serotype 51: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 51 | 5.70 (7.914)
  28-day dosing schedule: Week 48: Serotype 51: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 51 | 1.58 (0.843)
  21-day dosing schedule: Week 48: Serotype 51: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 51 | 5.86 (8.456)
  Baseline: Serotype 54 | 3.04 (4.819)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 54 | 2.33 (2.575)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 54 | 5.04 (6.363)
  28-day dosing schedule: Week 32: Serotype 54: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 54 | 2.95 (5.542)
  21-day dosing schedule: Week 30: Serotype 54: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 54 | 4.86 (5.637)
  28-day dosing schedule: Week 48: Serotype 54: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 54 | 2.53 (3.181)
  21-day dosing schedule: Week 48: Serotype 54: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 54 | 4.13 (3.700)
  Baseline: Serotype 56 | 3.41 (8.495)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 56 | 2.55 (6.989)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 56 | 5.84 (9.970)
  28-day dosing schedule: Week 32: Serotype 56: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 56 | 2.17 (5.089)
  21-day dosing schedule: Week 30: Serotype 56: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 56 | 5.38 (8.242)
  28-day dosing schedule: Week 48: Serotype 56: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 56 | 2.54 (8.116)
  21-day dosing schedule: Week 48: Serotype 56: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 56 | 6.00 (10.338)
  Baseline: Serotype 57 | 5.73 (8.398)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 57 | 5.11 (8.435)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 57 | 23.40 (48.403)
  28-day dosing schedule: Week 32: Serotype 57: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 57 | 5.46 (9.059)
  21-day dosing schedule: Week 30: Serotype 57: number analyzed (Participants) | 7
  21-day dosing schedule: Week 30: Serotype 57 | 7.00 (10.268)
  28-day dosing schedule: Week 48: Serotype 57: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 57 | 5.31 (9.379)
  21-day dosing schedule: Week 48: Serotype 57: number analyzed (Participants) | 7
  21-day dosing schedule: Week 48: Serotype 57 | 8.17 (12.789)
  Baseline: Serotype 68 | 1.08 (1.095)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 68 | 0.86 (0.567)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 68 | 1.66 (1.555)
  28-day dosing schedule: Week 32: Serotype 68: number analyzed (Participants) | 38
  28-day dosing schedule: Week 32: Serotype 68 | 0.93 (0.918)
  21-day dosing schedule: Week 30: Serotype 68: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 68 | 1.36 (1.260)
  28-day dosing schedule: Week 48: Serotype 68: number analyzed (Participants) | 38
  28-day dosing schedule: Week 48: Serotype 68 | 0.76 (0.524)
  21-day dosing schedule: Week 48: Serotype 68: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 68 | 1.33 (1.233)
  Baseline: Serotype 70 | 1.98 (2.911)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 70 | 1.43 (1.100)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 70 | 3.56 (5.360)
  28-day dosing schedule: Week 32: Serotype 70: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 70 | 1.53 (1.128)
  21-day dosing schedule: Week 30: Serotype 70: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 70 | 3.53 (5.776)
  28-day dosing schedule: Week 48: Serotype 70: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 70 | 1.48 (0.988)
  21-day dosing schedule: Week 48: Serotype 70: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 70 | 3.19 (3.978)
  Baseline: Serotype 8 | 2.10 (2.650)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 8 | 1.67 (1.258)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 8 | 3.51 (3.440)
  28-day dosing schedule: Week 32: Serotype 8: number analyzed (Participants) | 39
  28-day dosing schedule: Week 32: Serotype 8 | 1.86 (1.822)
  21-day dosing schedule: Week 30: Serotype 8: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 8 | 3.66 (4.268)
  28-day dosing schedule: Week 48: Serotype 8: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 8 | 1.82 (1.593)
  21-day dosing schedule: Week 48: Serotype 8: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 8 | 3.63 (3.479)
  Baseline: Serotype 9 | 0.96 (0.694)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16: Serotype 9 | 0.77 (0.510)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18: Serotype 9 | 1.03 (0.560)
  28-day dosing schedule: Week 32: Serotype 9: number analyzed (Participants) | 38
  28-day dosing schedule: Week 32: Serotype 9 | 0.81 (0.587)
  21-day dosing schedule: Week 30: Serotype 9: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30: Serotype 9 | 0.99 (0.503)
  28-day dosing schedule: Week 48: Serotype 9: number analyzed (Participants) | 39
  28-day dosing schedule: Week 48: Serotype 9 | 0.75 (0.433)
  21-day dosing schedule: Week 48: Serotype 9: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48: Serotype 9 | 1.03 (0.486)

7. Secondary Outcome: Anti-Measles Antibody Levels
Description: The anti-measles antibody levels were collected and analyzed at a central laboratory.
Time Frame: Baseline, Weeks 16, 32 and 48 (28-day dosing schedule); Weeks 18, 30, 48 (21-day dosing schedule)
Population: As per change in planned analysis, the anti-measles antibody level test was not performed.
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 0

8. Secondary Outcome: Anti-Haemophilus Influenza Type B Antibody Levels
Description: The anti-haemophilus influenza type B antibody levels were collected and analyzed at central laboratory.
Time Frame: Baseline, Weeks 16, 32 and 48 (28 -day dosing schedule); Weeks 18, 30, 48 (21-day dosing schedule)
Population: FAS included all participants who had received at least 1 dose of study medication. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per the dosing schedule.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
micrograms per milliliter (mcg/mL)
  Baseline | 2.010 (1.1641)
  28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16 | 2.547 (1.7879)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18 | 2.489 (0.9027)
  28-day dosing schedule: Week 32: number analyzed (Participants) | 38
  28-day dosing schedule: Week 32 | 2.277 (1.3112)
  21-day dosing schedule: Week 30: number analyzed (Participants) | 8
  21-day dosing schedule: Week 30 | 2.888 (0.8676)
  28-day dosing schedule: Week 48: number analyzed (Participants) | 35
  28-day dosing schedule: Week 48 | 2.183 (1.1944)
  21-day dosing schedule: Week 48: number analyzed (Participants) | 8
  21-day dosing schedule: Week 48 | 2.606 (0.8433)

9. Secondary Outcome: Incidence Rate of Any Infection Other Than Acute Serious Bacterial Infections
Description: Incidence rate was defined as the mean number of any infection other than acute serious bacterial infections (bacterial pneumonia, bacteraemia/sepsis, bacterial meningitis, visceral abscess, osteomyelitis/septic arthritis) per participant-year. Incidence rate of any infection other than acute bacterial serious infections collected by the participant/participants parent(s)/legal guardian(s) in the participant diary or during clinic visit was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who received at least 1 dose of study medication. Here, "Number Analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: infections per participant year
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
infections per participant year
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 4.2 (2.05)
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 1.6 (1.25)

10. Secondary Outcome: Duration of Any Infection Other Than Acute Serious Bacterial Infections
Description: Duration of any infection other than serious acute bacterial infections (in days) was calculated as date of stop of infection - date of start of infection + 1. Duration of any infection other than serious acute bacterial infections collected by the by the participant/participants parent(s)/legal guardian(s) in the participant diary or during clinic visit was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
days
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 42.9 (66.66)
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 25.3 (52.14)

11. Secondary Outcome: Incidence Rate of Fever Episodes
Description: Incidence rate was defined as the mean number of fever episodes per participant-year. Incidence rate of fever episodes collected by the participant/participant's parent(s)/legal guardian(s) in the participant diary or during clinic visit were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: fever episodes per participant year
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
fever episodes per participant year
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 0.0 (0.0)
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 0.2 (0.42)

12. Secondary Outcome: Duration of Fever Episodes in Participants
Description: Duration of fever episodes in participants was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who had fever episodes and "Number Analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 7
days
  21-day dosing schedule: number analyzed (Participants) | 0
  28-day dosing schedule | 3.0 (2.24)

13. Secondary Outcome: Duration of Overall Participants Hospitalization
Description: Duration of overall participants hospitalization was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who received at least 1 dose of study. Here, "Overall Number of Participants Analyzed" signifies those participants who were hospitalized and "Number Analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 4
days
  21-day dosing schedule: number analyzed (Participants) | 1
  21-day dosing schedule | 6.0
  28-day dosing schedule: number analyzed (Participants) | 3
  28-day dosing schedule | 3.3 (1.53)

14. Secondary Outcome: Duration of Participants Hospitalization Due to Infection
Description: Duration of participants hospitalization due to infection was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who were hospitalized due to infection.
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 0

15. Secondary Outcome: Incidence Rate of Antibiotics Episodes for Treatment of Any Kind of Infections
Description: Incidence rate was defined as the mean number of antibiotics episodes per participant year. Incidence rate of participants on antibiotics for treatment of any kind of infections was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: antibiotics episodes/participant year
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
antibiotics episodes/participant year
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 3.8 (1.95)
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 2.1 (1.46)

16. Secondary Outcome: Duration of Participants on Antibiotics for Treatment of Any Kind of Infection
Description: Duration of participants on antibiotics for treatment of any kind of infection was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who took antibiotics to treat infections and "Number Analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 36
days
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 13.1 (5.72)
  28-day dosing schedule: number analyzed (Participants) | 28
  28-day dosing schedule | 13.3 (35.86)

17. Secondary Outcome: Duration of Missed School/Work/Other Major Activities Due to Infections
Description: Duration of missed school/work/other major activities due to infections was reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: FAS included all participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who had missed school/work/other major activities due to infections and, "Number Analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 9
days
  21-day dosing schedule: number analyzed (Participants) | 3
  21-day dosing schedule | 25.3 (25.11)
  28-day dosing schedule: number analyzed (Participants) | 6
  28-day dosing schedule | 4.7 (2.73)

18. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL) Score
Description: 23-item PedsQL generic core scales was a modular approach to measure health-related Quality of Life (QoL) in healthy children, adolescents and those with acute and chronic health conditions. The total scale score (23 items) consisted of Physical Health Summary Score (8 items) and Psychosocial Health SummaryScore (15 items). Physical health summary included Physical Functioning (8 items) and Psychosocial health summary score included Emotional Functioning (5 items), Social Functioning (5 items) and School Functioning (5 items). Items were scored on a 5 point Likert-type response scale: 0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; and 4=almost always a problem). Once scored, items were reverse scored and linearly transformed to a 0-100 scale, where higher scores indicated better QoL. The overall range for total PedsQL score (23 items) was 0 to 100, with higher score indicated better QoL. Data for 18-25 years and >25 years age group was reported.
Time Frame: Baseline, Week 24 (21-day dosing schedule and 28-day dosing schedule), Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: The FAS included all participants who received at least 1 dose of study medication. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
score on a scale
  Baseline (18 to 25 years): number analyzed (Participants) | 2
  Baseline (18 to 25 years) | 87.5 (16.14)
  21-day dosing schedule: Week 24 (18 to 25 years): number analyzed (Participants) | 1
  21-day dosing schedule: Week 24 (18 to 25 years) | 68.5
  21-day dosing schedule: Week 51 (18 to 25 years): number analyzed (Participants) | 1
  21-day dosing schedule: Week 51 (18 to 25 years) | 58.7
  28-day dosing schedule: Week 24 (18 to 25 years): number analyzed (Participants) | 1
  28-day dosing schedule: Week 24 (18 to 25 years) | 100.0
  28-day dosing schedule: Week 52 (18 to 25 years): number analyzed (Participants) | 1
  28-day dosing schedule: Week 52 (18 to 25 years) | 100.0
  Baseline (> 25 years): number analyzed (Participants) | 45
  Baseline (> 25 years) | 76.2 (16.53)
  21-day dosing schedule: Week 24 (> 25 years): number analyzed (Participants) | 7
  21-day dosing schedule: Week 24 (> 25 years) | 65.1 (15.92)
  21-day dosing schedule: Week 51 (> 25 years): number analyzed (Participants) | 7
  21-day dosing schedule: Week 51 (> 25 years) | 70.3 (18.93)
  28-day dosing schedule: Week 24 (> 25 years): number analyzed (Participants) | 38
  28-day dosing schedule: Week 24 (> 25 years) | 78.3 (17.02)
  28-day dosing schedule: Week 52 (> 25 years): number analyzed (Participants) | 38
  28-day dosing schedule: Week 52 (> 25 years) | 77.8 (18.42)

19. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life- threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAE was defined as an AE with an onset that occurs after receiving study drug. Any TEAE included participants with both serious and non-serious TEAEs.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: The SAF included all participants who had received at least 1 dose of study medication. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  Participants with TEAEs: 21-day dosing schedule:: number analyzed (Participants) | 8
  Participants with TEAEs: 21-day dosing schedule: | 8
  Participants with TEAEs: 28-day dosing schedule: number analyzed (Participants) | 39
  Participants with TEAEs: 28-day dosing schedule | 38
  Participants with Serious TEAEs: 21-day dosing schedule: number analyzed (Participants) | 8
  Participants with Serious TEAEs: 21-day dosing schedule | 1
  Participants with Serious TEAEs: 28-day dosing schedule: number analyzed (Participants) | 39
  Participants with Serious TEAEs: 28-day dosing schedule | 3

20. Secondary Outcome: Number of TEAEs and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. A SAE was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life- threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. A TEAE was defined as an AE with an onset that occurs after receiving study drug. Number of TEAEs and Serious TEAEs were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: The SAF included all participants who had received at least 1 dose of study medication. "Overall Number of Participants Analyzed" signifies those participants who had TEAEs and "Number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Number; unit: adverse events
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 46
adverse events
  TEAEs: 21-day dosing schedule: number analyzed (Participants) | 8
  TEAEs: 21-day dosing schedule | 79
  TEAEs: 28-day dosing schedule: number analyzed (Participants) | 38
  TEAEs: 28-day dosing schedule | 324
  Serious TEAEs: 21-day dosing schedule: number analyzed (Participants) | 1
  Serious TEAEs: 21-day dosing schedule | 1
  Serious TEAEs: 28-day dosing schedule: number analyzed (Participants) | 3
  Serious TEAEs: 28-day dosing schedule | 4

21. Secondary Outcome: Number of Drug Related Infusion Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. Number of drug related infusion AEs were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: The SAF included all participants who have received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants who had drug related infusion AEs and "Number Anlyazed" signifies those who were evaluable at specified time points as per dosing schedule.
Measure: Number; unit: adverse events
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 19
adverse events
  21-day dosing schedule: number analyzed (Participants) | 2
  21-day dosing schedule | 3
  28-day dosing schedule: number analyzed (Participants) | 17
  28-day dosing schedule | 60

22. Secondary Outcome: Percentage of Participants Who Experienced at Least One Drug Related Infusion Adverse Events (AEs)
Description: Percentage of participants who experienced at least one drug related infusion AEs were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: The SAF included all participants who have received at least 1 dose of study medication. Here, "Number Analyzed" signifies those participants who were evaluable at specified time points as per the dosing schedule.
Measure: Number; unit: percentage of participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
percentage of participants
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 25.0
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 43.6

23. Secondary Outcome: Number of Infusions With Decreased Infusion Rate Due to Adverse Events (AEs)
Description: Number of infusions with decreased infusion rate due to AEs were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: as for outcome 22
Measure: Count of Units; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Number analyzed (Infusions) | 643
Infusions
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule: number analyzed (Infusions) | 136
  21-day dosing schedule | 0
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule: number analyzed (Infusions) | 507
  28-day dosing schedule | 9

24. Secondary Outcome: Number of Infusions With One or More Infusion Associated Adverse Events (AEs)
Description: The number of infusions with one or more infusion associated AEs were reported collectively for 21 and 28-day dosing schedule up to Week 52.
Time Frame: Baseline up to Week 52
Population: The SAF included all participants who have received at least 1 dose of study medication.
Measure: Count of Units; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Number analyzed (Infusions) | 643
Infusions | 80

25. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital signs included body temperature, systolic and diastolic blood pressure, heart rate and weight. The systolic and diastolic blood pressure and pulse rate was measured after the participants have in a rested at least 3 minutes in seated position. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in vital signs were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: SAF included all participants who have received at least 1 dose of study medication. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per the dosing schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 0
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 0

26. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Physical Examinations
Description: Physical examination included the examination of general appearance, skin, neck, eyes, ears, nose, throat, cardiovascular assessment including rhythm, and presence of other cardiac abnormalities (for example gallops, murmurs, cardiomegaly), respiratory system, gastrointestinal system, genitourinary system and musculoskeletal system. Clinical significance was decided by the investigator. The number of participants with clinically significant changes from baseline in physical examination were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  21-day dosing schedule: number analyzed (Participants) | 8
  21-day dosing schedule | 0
  28-day dosing schedule: number analyzed (Participants) | 39
  28-day dosing schedule | 0

27. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory parameters included chemistry, hematology and urinalysis. Clinical significance was determined by the investigator. The number of participants with clinically significant changes from baseline in laboratory parameters were reported.
Time Frame: Baseline up to Week 51 (21-day dosing schedule) and Week 52 (28-day dosing schedule)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  Hematology: 21-day dosing schedule: number analyzed (Participants) | 8
  Hematology: 21-day dosing schedule | 3
  Hematology: 28-day dosing schedule: number analyzed (Participants) | 39
  Hematology: 28-day dosing schedule | 7
  Chemistry: 21-day dosing schedule: number analyzed (Participants) | 8
  Chemistry: 21-day dosing schedule | 1
  Chemistry: 28-day dosing schedule: number analyzed (Participants) | 39
  Chemistry: 28-day dosing schedule | 5
  Urinalysis: 21-day dosing schedule: number analyzed (Participants) | 8
  Urinalysis: 21-day dosing schedule | 2
  Urinalysis: 28-day dosing schedule: number analyzed (Participants) | 39
  Urinalysis: 28-day dosing schedule | 4

28. Secondary Outcome: Number of Participants With Positive Coomb's Test at Week 16 (28-day Dosing Schedule) and Week 18 (21-day Dosing Schedule)
Description: Intravascular hemolysis testing was performed by using coomb's test. The coomb's assessment was performed at a central laboratory.
Time Frame: At Week 16 (28-day dosing schedule) and Week 18 (21-day dosing schedule)
Population: SAF included all participants who have received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies those participants with Coombs Test and "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 46
Participants
  28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16 | 14
  21-day dosing schedule: Week 18: number analyzed (Participants) | 7
  21-day dosing schedule: Week 18 | 4

29. Secondary Outcome: Number of Participants With Positive Urine Hemosiderin Test
Description: Number of participants with positive urine hemosiderin test were reported.
Time Frame: At Week 16 (28-day dosing schedule) and Week 18 (21-day dosing schedule)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16 | 0
  21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18 | 0

30. Secondary Outcome: Number of Participants With Abnormal Plasma-free Haemoglobin Level
Description: Number of participants with plasma-free haemoglobin level more than or equal to (>=) 69 milligrams per deciliter (mg/dL) were consisdered as abormal and were reported.
Time Frame: At Week 16 (28-day dosing schedule) and Week 18 (21-day dosing schedule)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16 | 10
  21-day dosing schedule : Week 18: number analyzed (Participants) | 8
  21-day dosing schedule : Week 18 | 2

31. Secondary Outcome: Number of Participants With Abnormal Serum Haptoglobin Level
Description: Number of participants with abnormal serum haptoglobin level were reported.
Time Frame: At Week 16 (28-day dosing schedule) and Week 18 (21-day dosing schedule)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 47
Participants
  28-day dosing schedule: Week 16: number analyzed (Participants) | 39
  28-day dosing schedule: Week 16 | 10
  21-day dosing schedule: Week 18: number analyzed (Participants) | 8
  21-day dosing schedule: Week 18 | 0

32. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Total Immunoglobulin G (IgG)
Description: Cmax was obtained directly from the concentration versus time curve. Both baseline corrected and un-corrected data was reported.
Time Frame: At Week 16 (28-day dosing schedule) and Week 18 (21-day dosing schedule), 10 to 30 minutes pre-infusion, 30 minutes, 2, 24, 72, 168, 336, 504, 672 hours post infusion
Population: Pharmacokinetic (PK) Evaluation Set: all adult participants that consent to this part of protocol and who have PK analysis performed at 5th infusion (28-day infusion schedule)/7th infusion (21-day infusion schedule). This set included all participants following principles of SAF for whom at least 1 concentration of total IgGs, IgG subclasses 1-4/IgG specific antibody levels. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
milligrams per deciliter (mg/dL)
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 1280 (433)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 1520 (185)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 2300 (466)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 2680 (282)

33. Secondary Outcome: Elimination Half-Life (t1/2) of Total IgG
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 was calculated by natural log 2 divided by Kel. Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: PK evaluation set was used. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
hours
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 158 (48.4)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 107 (45.4)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 896 (269)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 587 (58.2)

34. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of Total IgG
Description: Area under the serum concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: PK Evaluation Set: all adult participants that consent to this part of protocol and who have PK analysis performed at 5th infusion (28-day infusion schedule) or 7th infusion (21-day infusion schedule). This set included all participants following the principles of SAF for whom at least 1 concentration of total IgGs, IgG subclasses 1-4/IgG specific antibody levels. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: day*milligram per deciliter (day*mg/dL)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
day*milligram per deciliter (day*mg/dL)
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 9520 (3310)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 8380 (1670)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 37300 (7720)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 31700 (6030)

35. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Total IgG
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Kel, where Clast pred was the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above the Lower Limit of quantification (LLOQ) and Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hr*g/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 22
hr*g/L
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 2710.991 (733.1555)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline corrected: 21-day dosing schedule: Week 18 | 2435.562 (471.842)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 22065.3148 (5061.15798)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 18292.68 (2869.244)

36. Secondary Outcome: Area Under the Serum Concentration-Time Curve During a Dosing Interval (AUCtau) of Total IgG
Description: AUCtau was defined as area under the serum concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: day*mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
day*mg/dL
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 9840 (3330)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 8860 (1630)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 38000 (6500)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 34000 (3630)

37. Secondary Outcome: Volume of Distribution (Vd) of Total IgG
Description: Vd was defined as the the theoretical volume in which the total amount of total IgG would need to be uniformly distributed to produce the desired blood concentration of a total IgG. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: deciliters per kilogram (dL/kg)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
deciliters per kilogram (dL/kg)
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 0.532 (0.108)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 0.563 (0.161)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 0.697 (0.118)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 0.667 (0.0398)

38. Secondary Outcome: Steady State Clearance (CLss) of Total IgG
Description: Clearance of a total IgG was a measure of the rate at which a total IgG is metabolized or eliminated by normal biological processes. CLss of total IgG was measured in milliliters per hour per kilogram (mL/hr/kg). Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: dL/day/kg
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
dL/day/kg
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 0.0559 (0.0102)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 0.0763 (0.00342)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 0.0140 (0.00355)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 0.0193 (0.00305)

39. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Total IgG
Description: Cmin was minimum observed serum concentration obtained directly from the concentration versus time curve. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
mg/dL
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 0.00 (0.00)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 0.00 (0.00)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 994 (200)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 1140 (150)

40. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) of Total IgG
Description: Tmax was obtained directly from the concentration versus time curve. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Median (Full Range); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
hours
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 0.515 [0.500 to 23.8]
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 0.530 [0.500 to 2.02]
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 0.515 [0.500 to 23.8]
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 0.530 [0.500 to 2.02]

41. Secondary Outcome: Elimination Rate Constant (Kel) of Total IgG
Description: Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
1/hour
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 0.0048 (0.00156)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 0.00743 (0.00300)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 0.000845 (0.000270)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 0.00119 (0.000117)

42. Secondary Outcome: Average Concentration of Total IgG Over the Dosing Interval (Cavg)
Description: Average concentration of total IgG over the dosing interval (Cavg) was reported. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: PK Evaluation Set: all adult participants that consent to this part of protocol and who have PK analysis performed at 5th infusion (28-day infusion schedule)/7th infusion (21-day infusion schedule). This set included all participants following principles of SAF for whom at least 1 concentration of total IgGs, IgG subclasses 1-4/IgG specific antibody levels. Here, "number analyzed" signifies those participants who were evaluable at specified time points as per dosing schedule.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
mg/dL
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 354 (117)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 424 (78.6)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 1370 (239)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 1630 (175)

43. Secondary Outcome: Percentage Peak Trough Fluctuation of Total IgG
Description: The peak trough fluctuation within complete dosing interval at steady state of total IgG was reported. Both baseline corrected and un-corrected data was reported.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: percent fluctuation
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
percent fluctuation
  Baseline corrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline corrected: 28-day dosing schedule: Week 16 | 364 (70.7)
  Baseline corrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  Baseline corrected: 21-day dosing schedule: Week 18 | 360 (56.3)
  Baseline uncorrected: 28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  Baseline uncorrected: 28-day dosing schedule: Week 16 | 94.3 (30.6)
  Baseline uncorrected: 21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  Baseline uncorrected: 21-day dosing schedule: Week 18 | 95.0 (7.92)

44. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
IU/mL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16 | 6.533 (2.9955)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 7.400 (2.0988)

45. Secondary Outcome: Elimination Half-Life (t1/2) of Antigen-Specific Tetanus Toxoid Antibodies
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 was calculated by natural log 2 divided by Kel. Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
hours
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 618.97 (320.008)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 1097.75 (1061.343)

46. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Area under the serum concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule. The AUC0-t of antigen-specific tetanus toxoid antibodies was measured in hour*international units per milliliter (hr*IU/mL).
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: hr*IU/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
hr*IU/mL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16 | 2037.7497 (568.85079)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 1805.9758 (210.37005)

47. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Antigen-Specific Tetanus Toxoid Antibodies
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Kel, where Clast pred was the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above the Lower Limit of quantification (LLOQ) and Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter(hr*mcg/mL)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
hour*microgram per milliliter(hr*mcg/mL)
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 4171.4977 (2513.60199)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 10142.0162 (12855.54687)

48. Secondary Outcome: Area Under the Serum Concentration-Time Curve During a Dosing Interval (AUCtau) of Antigen-Specific Tetanus Toxoid Antibodies
Description: AUCtau was defined as area under the serum concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hr*IU/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
hr*IU/mL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 1997.8829 (526.07254)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 1934.6533 (317.07241)

49. Secondary Outcome: Volume of Distribution (Vd) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Vd was defined as the the theoretical volume in which the total amount of antigen-specific tetanus toxoid antibodies would need to be uniformly distributed to produce the desired blood concentration of antigen-specific tetanus toxoid antibodies. The Vd of antigen-specific tetanus toxoid antibodies was measured in milligrams*milliliter per international unit*kilogram (mg*mL/IU*kg).
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg*mL/IU*kg
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
mg*mL/IU*kg
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 263.3132 (157.80776)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 688.4792 (792.01235)

50. Secondary Outcome: Steady State Clearance (CLss) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Clearance of a antigen-specific tetanus toxoid antibodies was a measure of the rate at which a antigen-specific tetanus toxoid antibodies are metabolized or eliminated by normal biological processes. The CLss of antigen-specific tetanus toxoid antibodies was reported. The CLss of antigen-specific tetanus toxoid antibodies was measured in milligrams*milliliter per hour*international unit*kilogram (mg*mL/hr*IU*kg).
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg*mL/hr*IU*kg
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
mg*mL/hr*IU*kg
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 0.2741 (0.06916)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 0.3724 (0.05201)

51. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Cmin was minimum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
IU/mL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16 | 1.833 (0.5531)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 2.240 (0.4827)

52. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Median (Full Range); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
hours
  28-day dosing schedule: Week 16: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16 | 2.000 [0.48 to 168.00]
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 70.450 [1.97 to 71.25]

53. Secondary Outcome: Elimination Rate Constant (Kel) of Antigen-Specific Tetanus Toxoid Antibodies
Description: Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 11
1/hour
  28-day dosing schedule: Week 16: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16 | 0.0014 (0.00062)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 0.0011 (0.00065)

54. Secondary Outcome: Average Concentration of Antigen-Specific Tetanus Toxoid Antibodies Over the Dosing Interval (Cavg)
Description: Average concentration of antigen-specific tetanus toxoid antibodies over the dosing interval (Cavg) was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
IU/mL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 2.9730 (0.78285)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 3.8386 (0.62911)

55. Secondary Outcome: Percentage Peak Trough Fluctuation of Antigen-Specific Tetanus Toxoid Antibodies
Description: The peak trough fluctuation within complete dosing interval at steady state of antigen-specific tetanus toxoid antibodies was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percent fluctuation
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
percent fluctuation
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 154.7237 (63.56527)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 145.9127 (55.92179)

56. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 22
milligram per deciliter (mg/dL)
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 0.682 (0.204)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 0.787 (0.141)

57. Secondary Outcome: Elimination Half-Life (t1/2) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: as for outcome 45
Time Frame: as for outcome 32
Population: PK evaluation set was used. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable at specified time pointsas per dosing schedule.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 15
hours
  28-day dosing schedule: Week 16: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16 | 682 (488)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18 | 364 (52.2)

58. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Area under the serum concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule. AUC0-t of antigen-specific haemophilus influenza Type B Antibodies was measured in hour*microgram per milliliter (hr*mcg/mL).
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: day*mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 22
day*mg/dL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 9.80 (4.35)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 8.80 (3.02)

59. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: as for outcome 47
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 20
hr*mcg/mL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 5087.4141 (3563.09258)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18 | 4223.1698 (493.35835)

60. Secondary Outcome: Area Under the Serum Concentration-Time Curve During a Dosing Interval (AUCtau) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: as for outcome 48
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: day*mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
day*mg/dL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 9.80 (4.35)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 9.90 (2.03)

61. Secondary Outcome: Volume of Distribution (Vd) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Vd was defined as the the theoretical volume in which the total amount of antigen-specific haemophilus influenza type B antibodies would need to be uniformly distributed to produce the desired blood concentration of a antigen-specific haemophilus influenza type B antibodies.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: milligrams per kilogram (mL/kg)
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 20
milligrams per kilogram (mL/kg)
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 245966.4231 (160457.69395)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18 | 182273.0408 (88143.84190)

62. Secondary Outcome: Steady State Clearance (CLss) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Clearance of antigen-specific haemophilus influenza type B antibodies was a measure of the rate at which antigen-specific haemophilus influenza type B antibodies were metabolized or eliminated by normal biological processes. CLss of antigen-specific haemophilus influenza type B antibodies was measured in milliliter per hour per kilogram (mL/hr/kg).
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 20
mL/hr/kg
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 253.5539 (75.88763)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18 | 299.5030 (100.44087)

63. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Cmin was minimum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 22
mg/dL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 0.215 (0.134)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 0.225 (0.0623)

64. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Median (Full Range); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 22
hours
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 0.500 [0.480 to 24.3]
  21-day dosing schedule: Week 18: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 | 2.02 [0.500 to 502]

65. Secondary Outcome: Terminal Elimination Rate Constant (Lambda z) of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: Terminal Elimination Rate Constant (lambda z) derived if data allowed based on PK acceptance criteria
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 15
1/hour
  28-day dosing schedule: Week 16: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16 | 0.00148 (0.000815)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18 | 0.00192 (0.000276)

66. Secondary Outcome: Average Concentration of Antigen-Specific Haemophilus Influenza Type B Antibodies Over the Dosing Interval (Cavg)
Description: Average concentration of antigen-specific haemophilus influenza type B antibodies over the dosing interval (Cavg) was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
mg/dL
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 0.352 (0.155)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 0.474 (0.0971)

67. Secondary Outcome: Percentage Peak Trough Fluctuation of Antigen-Specific Haemophilus Influenza Type B Antibodies
Description: The peak trough fluctuation within complete dosing interval at steady state of antigen-specific haemophilus influenza type B antibodies was reported.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percent fluctuation
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
percent fluctuation
  28-day dosing schedule: Week 16: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16 | 141 (72.8)
  21-day dosing schedule: Week 18: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18 | 88.1 (66.9)

68. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: Cmax was obtained directly from the concentration versus time curve. The Cmax for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8, serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
mg/L
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 1 | 3.478 (2.7623)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 12 | 1.256 (1.2458)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 14 | 20.378 (46.3772)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 17 | 4.350 (5.6783)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 19 | 7.767 (8.5255)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 2 | 3.822 (1.2758)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 20 | 4.728 (3.0665)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 22 | 2.050 (1.3382)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 23 | 3.039 (3.3482)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 26 | 2.433 (1.3569)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 3 | 2.933 (1.6150)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 0.685 (0.2410)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 34 | 2.472 (0.9940)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 43 | 2.572 (1.1108)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 5 | 5.217 (4.0965)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 51 | 3.611 (1.3788)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 54 | 4.806 (2.0783)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 56 | 5.778 (11.7004)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 57 | 12.511 (21.4792)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 68 | 1.806 (0.8033)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 70 | 3.228 (1.6080)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 8 | 3.683 (2.6600)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 9 | 1.583 (0.7148)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 1 | 8.440 (8.3182)
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 12 | 1.140 (0.1673)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 14 | 11.280 (3.5053)
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 17 | 5.860 (4.0930)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 19 | 6.440 (1.0691)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 2 | 6.180 (4.6370)
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 20 | 5.580 (1.8754)
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 22 | 4.420 (5.4422)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 23 | 2.360 (0.8620)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 26 | 3.340 (2.5373)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 3 | 9.720 (12.7874)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 34 | 5.060 (6.2843)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 4 | 0.980 (0.6301)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 43 | 2.660 (0.7403)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 5 | 10.160 (12.4969)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 51 | 11.700 (14.2886)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 54 | 9.820 (10.6338)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 56 | 13.300 (19.3380)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 57 | 5.825 (0.9878)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 68 | 2.460 (1.7009)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 70 | 6.260 (7.0741)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 8 | 6.120 (4.5510)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 9 | 1.980 (0.7294)

69. Secondary Outcome: Elimination Half-Life (t1/2) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: t1/2 was the time measured for the concentration to decrease by one half. t1/2 was calculated by natural log 2 divided by Kel. Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase.Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. The t1/2 for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 13
hours
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 1 | 533.06 (279.860)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 12 | 415.27 (104.179)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 14 | 737.33 (293.005)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 17 | 568.11 (184.079)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 19 | 794.76 (365.625)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 5
  28-day dosing schedule: Week 16: Serotype 2 | 943.63 (597.812)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 20 | 977.87 (511.568)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 22 | 574.22 (258.366)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 23 | 837.29 (476.321)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 26 | 638.60 (285.966)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 10
  28-day dosing schedule: Week 16: Serotype 3 | 626.69 (275.200)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 34 | 680.14 (400.291)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 3
  28-day dosing schedule: Week 16: Serotype 4 | 522.15 (39.466)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 9
  28-day dosing schedule: Week 16: Serotype 43 | 573.32 (191.776)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 5 | 632.03 (220.955)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 51 | 794.63 (474.015)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 54 | 1184.97 (1088.054)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 56 | 527.75 (144.729)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 57 | 1346.21 (1574.359)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 68 | 688.31 (354.982)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 9
  28-day dosing schedule: Week 16: Serotype 70 | 709.41 (282.061)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 8 | 562.30 (138.178)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 4
  28-day dosing schedule: Week 16: Serotype 9 | 555.66 (274.555)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 1 | 813.74
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 12 | 498.21 (105.271)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 14 | 1467.24
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 17 | 1161.62 (409.606)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 19 | 839.73 (867.812)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 2 | 860.60
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 20 | 779.88
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 22 | 966.61 (104.462)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 23 | 805.76 (155.609)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 26 | 900.44
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 3 | 292.95
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 34 | 820.04 (92.314)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 4 | 638.35 (549.756)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 43 | 295.34 (120.334)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 5 | 825.99
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 51 | 813.32
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 54 | 754.20
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 56 | 931.50
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 68 | 259.63
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 70 | 1437.71 (1083.055)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 8 | 616.54
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 9 | 890.30

70. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: Area under the serum concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule. AUC0-t of antigen-pneumococcal capsular polysaccharide was measured in hour*microgram per milliliter (hr*mcg/mL). The AUC0-t for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: hr*mg/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
hr*mg/L
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 1 | 1267.2703 (1231.86109)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 12 | 481.8080 (615.13837)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 14 | 7680.6757 (17443.37339)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 17 | 1707.2987 (2326.27590)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 19 | 3264.5178 (4922.67289)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 2 | 1462.1037 (491.94211)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 20 | 1776.5915 (1472.71297)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 22 | 767.3831 (752.08067)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 23 | 1206.7604 (1547.47617)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 26 | 929.6216 (696.05624)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 3 | 940.1352 (397.58653)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 34 | 916.8877 (339.74807)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 245.8296 (89.81281)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 43 | 901.9934 (415.28147)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 5 | 1882.0174 (1606.54653)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 51 | 1313.1756 (285.57756)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 54 | 1659.0010 (487.17054)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 56 | 2361.1009 (5435.67901)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 57 | 5140.5242 (10426.05050)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 68 | 637.6826 (180.23219)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 70 | 1239.3842 (746.05163)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 8 | 1396.1732 (1343.80361)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 9 | 545.3315 (201.37388)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 1 | 3361.3444 (3529.24121)
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 12 | 364.7574 (66.07380)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 14 | 4026.2582 (1827.76472)
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 17 | 2327.4433 (1869.77732)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 19 | 2139.8818 (546.99394)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 2 | 2388.1819 (2054.90148)
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 20 | 2088.0431 (956.15600)
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 22 | 1728.1721 (2363.07921)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 23 | 826.4154 (390.75602)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 26 | 1199.7678 (1115.65007)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 3 | 3834.6179 (5425.47048)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 34 | 2095.6088 (2982.98719)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 4 | 363.5605 (289.99268)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 43 | 919.1971 (290.08829)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 5 | 4050.8597 (5582.10279)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 51 | 4775.1477 (6034.17097)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 54 | 3849.0042 (4696.54103)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 56 | 5069.9328 (7483.01937)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 57 | 1946.7526 (134.44174)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 68 | 900.2735 (757.57732)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 70 | 2385.0419 (3013.20369)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 8 | 2555.3317 (2162.87976)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 9 | 707.9849 (310.25117)

71. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: AUC0-inf was calculated by combining AUC0-t and AUCextra. AUCextra represents an extrapolated value obtained by Clast pred/Kel, where Clast pred was the calculated serum concentration at the last sampling time point at which the measured serum concentration is at or above the Lower Limit of quantification (LLOQ) and Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. The AUC0-inf for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20 serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hr*mg/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 3
hr*mg/L
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 1 | 835.7493
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 17 | 815.5984
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 2
  28-day dosing schedule: Week 16: Serotype 22 | 706.0824 (101.30543)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 3 | 753.3039
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 56 | 871.0663
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 9 | 494.5129
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 43 | 1072.8342
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 0

72. Secondary Outcome: Area Under the Serum Concentration-Time Curve During a Dosing Interval (AUCtau) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: AUCtau was defined as area under the serum concentration-time curve from time zero to the end of the dosing interval (tau). AUCtau was calculated using the mixed log linear trapezoidal rule. The AUCtau for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: hr*mg/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
hr*mg/L
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 1 | 1295.2208 (1284.98717)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 12 | 496.5246 (652.01919)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 14 | 7938.1617 (18005.53693)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 17 | 1128.6509 (606.69308)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 19 | 2051.7286 (805.43957)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 2 | 1437.7169 (551.52102)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 20 | 1738.1297 (1558.89268)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 22 | 759.1847 (785.00558)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 23 | 1221.7947 (1608.36169)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 26 | 929.6706 (739.10055)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 3 | 902.9745 (415.50944)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 34 | 879.5261 (347.31703)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 241.3102 (93.08585)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 43 | 934.7032 (507.01946)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 15
  28-day dosing schedule: Week 16: Serotype 5 | 1525.6893 (617.53144)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 51 | 1327.8807 (304.68999)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 54 | 1665.6043 (473.20463)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 56 | 2456.3187 (5608.60157)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 57 | 5157.6297 (10068.88936)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 68 | 646.0577 (303.83828)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 70 | 1242.0569 (791.72945)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 15
  28-day dosing schedule: Week 16: Serotype 8 | 1112.3875 (364.77366)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 9 | 549.2854 (205.21945)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 1 | 3427.1894 (4395.22135)
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 12 | 340.6625 (40.16239)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 14 | 4203.7328 (2074.59529)
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 17 | 2120.4069 (1774.61729)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 19 | 2588.0431 (884.21458)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 2 | 1995.4796 (1312.64625)
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 20 | 2571.9984 (1782.65587)
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 22 | 860.7046 (377.70459)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 23 | 1074.8702 (591.84867)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 26 | 1640.1471 (1585.98684)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 3 | 6340.4080 (9208.98601)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 34 | 871.0315 (46.94825)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 4 | 464.1417 (438.74819)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 43 | 971.2482 (311.33350)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 5 | 1536.7299 (239.98044)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 51 | 5984.7197 (8063.82766)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 54 | 4422.4410 (5245.59189)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 56 | 6780.9969 (9967.85603)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 57 | 2280.6541 (245.58661)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 68 | 1209.1992 (1169.34365)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 70 | 1136.7545 (243.27839)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 8 | 2145.6232 (1950.12455)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 9 | 764.0375 (331.36438)

73. Secondary Outcome: Volume of Distribution (Vd) of of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: Vd was defined as the the theoretical volume in which the total amount of anti-pneumococcal capsular polysaccharide would need to be uniformly distributed to produce the desired blood concentration of a anti-pneumococcal capsular polysaccharide. The Vd for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 3
mL/kg
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 1 | 329057.3200
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 17 | 341197.1700
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 2
  28-day dosing schedule: Week 16: Serotype 22 | 231539.8050 (104298.38458)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 3 | 226738.9500
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 56 | 342896.0600
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 9 | 526016.9000
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 43 | 283171.4700
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 0

74. Secondary Outcome: Steady State Clearance (CLss) of Anti-pneumococcal Capsular Polysaccharide Antibodies (Overall SP Serotypes)
Description: Clearance of a anti-pneumococcal capsular polysaccharide antibodies was a measure of the rate at which a anti-pneumococcal capsular polysaccharide antibodies are metabolized or eliminated by normal biological processes. The CLss of anti-pneumococcal capsular polysaccharide antibodies was reported. The CLss of anti-pneumococcal capsular polysaccharide antibodies was measured in milligrams*milliliter per hour*international unit*kilogram (mg*mL/hr*IU*kg). The CLss for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg*mL/hr*IU*kg
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 3
mg*mL/hr*IU*kg
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 1 | 860.4600
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 17 | 862.3000
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 2
  28-day dosing schedule: Week 16: Serotype 22 | 604.0850 (190.31779)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 3 | 705.5700
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 56 | 854.8300
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 0
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 1
  28-day dosing schedule: Week 16: Serotype 9 | 1441.7300
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 43 | 849.0400
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 0

75. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: Cmin was minimum observed serum concentration obtained directly from the concentration versus time curve. The Cmin for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
mg/L
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 1 | 1.167 (0.7577)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 12 | 0.528 (0.8259)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 14 | 8.361 (19.9012)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 17 | 2.328 (4.4311)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 19 | 3.783 (6.2568)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 2 | 1.656 (0.8487)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 20 | 1.689 (0.7522)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 22 | 0.817 (1.0257)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 23 | 1.228 (1.8588)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 26 | 0.978 (0.6804)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 3 | 0.950 (0.5924)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 34 | 1.033 (0.6903)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 0.277 (0.1235)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 43 | 0.983 (0.6600)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 5 | 2.306 (3.2598)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 51 | 1.406 (0.4771)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 54 | 1.733 (0.6598)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 56 | 2.750 (6.7280)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 57 | 5.422 (10.7795)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 68 | 0.728 (0.4390)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 70 | 1.350 (0.9931)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 8 | 1.294 (0.6476)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 9 | 0.517 (0.2550)
  21-day dosing schedule: Week 18 : Serotype 1: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 1 | 5.400 (6.4211)
  21-day dosing schedule: Week 18 : Serotype 12: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 12 | 0.440 (0.1817)
  21-day dosing schedule: Week 18 : Serotype 14: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 14 | 5.880 (4.0084)
  21-day dosing schedule: Week 18 : Serotype 17: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 17 | 3.700 (3.3978)
  21-day dosing schedule: Week 18 : Serotype 19: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 19 | 2.940 (1.3107)
  21-day dosing schedule: Week 18 : Serotype 2: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 2 | 3.600 (3.6159)
  21-day dosing schedule: Week 18 : Serotype 20: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 20 | 3.120 (1.8992)
  21-day dosing schedule: Week 18 : Serotype 22: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 22 | 2.520 (3.6486)
  21-day dosing schedule: Week 18 : Serotype 23: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 : Serotype 23 | 1.200 (0.8660)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 26 | 1.740 (1.9191)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 3 | 5.920 (8.6126)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 34 | 3.220 (5.0226)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 4 | 0.520 (0.5630)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 43 | 1.300 (0.8031)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 5 | 6.240 (9.6619)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 51 | 7.620 (10.4406)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 54 | 5.980 (8.1515)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 56 | 7.820 (12.0038)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 57 | 2.375 (0.5909)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 68 | 1.400 (1.5700)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 70 | 3.920 (5.6971)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 8 | 4.260 (4.2846)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 9 | 1.040 (0.6804)

76. Secondary Outcome: Time to Reach the Maximum Serum Concentration (Tmax) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: Tmax was obtained directly from the concentration versus time curve. The Tmax for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 34
Measure: Median (Full Range); unit: hours
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 23
hours
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 1 | 0.542 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 12 | 0.517 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 14 | 1.417 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 17 | 1.992 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 19 | 0.642 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 2 | 1.458 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 22 | 0.500 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 23 | 0.642 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 26 | 0.642 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 3 | 0.517 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 34 | 1.758 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 0.500 [0.48 to 24.10]
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 43 | 1.750 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 5 | 0.642 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 51 | 0.650 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 54 | 0.642 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 56 | 1.633 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 57 | 0.642 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 68 | 0.650 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 70 | 0.500 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 8 | 0.542 [0.48 to 529.75]
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 9 | 0.500 [0.48 to 529.75]
  21-day dosing schedule: Week 18 Serotype 1: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 Serotype 1 | 71.250 [1.78 to 334.37]
  21-day dosing schedule: Week 18 Serotype 12: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 Serotype 12 | 1.783 [0.50 to 334.37]
  21-day dosing schedule: Week 18 Serotype 14: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18 Serotype 14 | 70.450 [0.50 to 334.37]
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 17 | 71.250 [1.78 to 337.30]
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 19 | 1.967 [0.53 to 334.37]
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 2 | 71.250 [1.78 to 337.30]
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 20 | 2.050 [1.78 to 457.00]
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 22 | 71.250 [1.78 to 337.30]
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 23 | 2.050 [0.50 to 334.37]
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 26 | 71.250 [1.78 to 334.37]
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 3 | 71.250 [2.05 to 457.00]
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 34 | 1.967 [0.53 to 334.37]
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 4 | 1.783 [0.50 to 334.37]
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 43 | 1.967 [0.53 to 457.00]
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 5 | 71.250 [1.78 to 337.30]
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 51 | 71.250 [0.53 to 334.37]
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 54 | 71.250 [1.78 to 334.37]
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 56 | 71.250 [1.78 to 334.37]
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 57 | 70.850 [0.53 to 334.37]
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 68 | 24.700 [0.50 to 334.37]
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 70 | 1.967 [0.48 to 71.25]
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 8 | 2.050 [1.78 to 334.37]
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 5
  21-day dosing schedule: Week 18: Serotype 9 | 70.450 [0.53 to 334.37]

77. Secondary Outcome: Elimination Rate Constant (Kel) of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: Kel was the elimination rate constant determined by log-linear regression analysis of the measured serum concentrations of the terminal log-linear phase. The Kel for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20 serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 12
1/hour
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 1 | 0.0016 (0.00081)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 12 | 0.0017 (0.00037)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 14 | 0.0011 (0.00037)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 17 | 0.0014 (0.00069)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 19 | 0.0010 (0.00039)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 5
  28-day dosing schedule: Week 16: Serotype 2 | 0.0010 (0.00054)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 20 | 0.0009 (0.00063)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 22 | 0.0015 (0.00082)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 23 | 0.0010 (0.00038)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 26 | 0.0013 (0.00057)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 10
  28-day dosing schedule: Week 16: Serotype 3 | 0.0014 (0.00078)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 34 | 0.0013 (0.00068)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 3
  28-day dosing schedule: Week 16: Serotype 4 | 0.0013 (0.00011)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 9
  28-day dosing schedule: Week 16: Serotype 43 | 0.0013 (0.00041)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 5 | 0.0012 (0.00036)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 51 | 0.0012 (0.00072)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 54 | 0.0009 (0.00052)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 56 | 0.0014 (0.00053)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 8
  28-day dosing schedule: Week 16: Serotype 57 | 0.0010 (0.00059)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 6
  28-day dosing schedule: Week 16: Serotype 68 | 0.0012 (0.00051)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 9
  28-day dosing schedule: Week 16: Serotype 70 | 0.0011 (0.00047)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 7
  28-day dosing schedule: Week 16: Serotype 8 | 0.0013 (0.00043)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 4
  28-day dosing schedule: Week 16: Serotype 9 | 0.0015 (0.00083)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 1 | 0.0009
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 12 | 0.0014 (0.00030)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 14 | 0.0005
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 17 | 0.0006 (0.00022)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 19 | 0.0018 (0.00183)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 2 | 0.0008
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 20 | 0.0009
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 22 | 0.0007 (0.00008)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 23 | 0.0009 (0.00017)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 26 | 0.0008
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 3 | 0.0024
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 34 | 0.0009 (0.00010)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 4 | 0.0016 (0.00094)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 43 | 0.0026 (0.00104)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 5 | 0.0008
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 51 | 0.0009
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 54 | 0.0009
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 56 | 0.0007
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 0
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 68 | 0.0027
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 2
  21-day dosing schedule: Week 18: Serotype 70 | 0.0007 (0.00051)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 8 | 0.0011
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 1
  21-day dosing schedule: Week 18: Serotype 9 | 0.0008

78. Secondary Outcome: Average Concentration of Anti-pneumococcal Capsular Polysaccharide the Dosing Interval (Cavg) (Overall SP Serotypes)
Description: Average concentration of anti-pneumococcal capsular polysaccharide over the dosing interval (Cavg) was reported. The Cavg for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 21
mg/L
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 1 | 1.9274 (1.91218)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 12 | 0.7389 (0.97027)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 14 | 11.8127 (26.793)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 17 | 1.7723 (0.86237)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 19 | 3.2992 (1.55795)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 2 | 2.2719 (0.84758)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 20 | 2.6925 (2.27169)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 22 | 1.1703 (1.14923)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 23 | 1.8608 (2.37096)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 26 | 1.4473 (1.09160)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 3 | 1.4018 (0.57076)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 34 | 1.4310 (0.67369)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 0.3715 (0.13038)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 43 | 1.3909 (0.75449)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 15
  28-day dosing schedule: Week 16: Serotype 5 | 2.2704 (0.91895)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 51 | 1.9760 (0.45341)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 54 | 2.4786 (0.70417)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 56 | 3.6552 (8.34613)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 57 | 7.7851 (14.9518)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 68 | 1.0037 (0.43741)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 70 | 1.8656 (1.16519)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 15
  28-day dosing schedule: Week 16: Serotype 8 | 1.6553 (0.54282)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 9 | 0.8174 (0.30539)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 1 | 6.8000 (8.72068)
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 12 | 0.6759 (0.07969)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 14 | 8.3407 (4.11626)
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 17 | 3.3332 (2.49783)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 19 | 4.1177 (1.24514)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 2 | 3.1566 (1.78858)
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 20 | 4.0521 (2.44372)
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 22 | 1.3653 (0.45325)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 23 | 1.6720 (0.80975)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 26 | 2.5183 (2.29821)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 3 | 9.6039 (13.55999)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 34 | 1.4352 (0.21030)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 4 | 0.7559 (0.61634)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 43 | 1.9271 (0.61773)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 5 | 3.0491 (0.47615)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 51 | 11.8744 (15.99966)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 54 | 8.7747 (10.40792)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 56 | 13.4544 (19.77749)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 57 | 3.7348 (0.38721)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 68 | 1.8682 (1.69358)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 70 | 2.0323 (0.31507)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 8 | 4.2572 (3.86929)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 9 | 1.5159 (0.65747)

79. Secondary Outcome: Percentage Peak Trough Fluctuation of Anti-pneumococcal Capsular Polysaccharide (Overall SP Serotypes)
Description: The peak trough fluctuation within complete dosing interval at steady state of anti-pneumococcal capsular polysaccharide was reported. The peak trough fluctuation for serotype 1, serotype 12, serotype 14, serotype 17, serotype 19, serotype 2, serotype 20, serotype 22, serotype 23, serotype 26, serotype 3, serotype 4, serotype 34, serotype 43, serotype 5, serotype 51, serotype 54, serotype 56, serotype 57, serotype 68, serotype 70, serotype 8 and serotype 9 was reported at Week 16 during 28-day dosing schedule and at Week 18 during 21-day dosing schedule.
Time Frame: as for outcome 32
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percent fluctuation
Arm/Group | Kedrion IVIG 10%
Number analyzed (Participants) | 22
percent fluctuation
  28-day dosing schedule: Week 16: Serotype 1: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 1 | 128.3177 (62.60668)
  28-day dosing schedule: Week 16: Serotype 12: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 12 | 125.2166 (64.54247)
  28-day dosing schedule: Week 16: Serotype 14: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 14 | 107.5731 (40.60933)
  28-day dosing schedule: Week 16: Serotype 17: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 17 | 103.6118 (35.89546)
  28-day dosing schedule: Week 16: Serotype 19: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 19 | 110.9054 (50.44522)
  28-day dosing schedule: Week 16: Serotype 2: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 2 | 105.2306 (55.00248)
  28-day dosing schedule: Week 16: Serotype 20: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 20 | 114.6004 (41.03380)
  28-day dosing schedule: Week 16: Serotype 22: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 22 | 128.1639 (58.30342)
  28-day dosing schedule: Week 16: Serotype 23: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 23 | 116.7754 (45.77432)
  28-day dosing schedule: Week 16: Serotype 26: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 26 | 122.7546 (65.89653)
  28-day dosing schedule: Week 16: Serotype 3: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 3 | 139.1737 (50.45738)
  28-day dosing schedule: Week 16: Serotype 34: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 34 | 112.0465 (48.26345)
  28-day dosing schedule: Week 16: Serotype 4: number analyzed (Participants) | 13
  28-day dosing schedule: Week 16: Serotype 4 | 117.2909 (65.62829)
  28-day dosing schedule: Week 16: Serotype 43: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 43 | 125.0358 (49.91946)
  28-day dosing schedule: Week 16: Serotype 5: number analyzed (Participants) | 15
  28-day dosing schedule: Week 16: Serotype 5 | 124.7428 (49.15063)
  28-day dosing schedule: Week 16: Serotype 51: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 51 | 110.9231 (48.65621)
  28-day dosing schedule: Week 16: Serotype 54: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 54 | 123.3022 (53.42626)
  28-day dosing schedule: Week 16: Serotype 56: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 56 | 116.6480 (52.81535)
  28-day dosing schedule: Week 16: Serotype 57: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 57 | 111.5242 (42.65179)
  28-day dosing schedule: Week 16: Serotype 68: number analyzed (Participants) | 16
  28-day dosing schedule: Week 16: Serotype 68 | 114.0701 (58.01418)
  28-day dosing schedule: Week 16: Serotype 70: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 70 | 109.4081 (43.80010)
  28-day dosing schedule: Week 16: Serotype 8: number analyzed (Participants) | 18
  28-day dosing schedule: Week 16: Serotype 8 | 117.3221 (38.97972)
  28-day dosing schedule: Week 16: Serotype 9: number analyzed (Participants) | 17
  28-day dosing schedule: Week 16: Serotype 9 | 130.6095 (65.79680)
  21-day dosing schedule: Week 18: Serotype 1: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 1 | 81.4603 (40.27141)
  21-day dosing schedule: Week 18: Serotype 12: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 12 | 102.9813 (10.00904)
  21-day dosing schedule: Week 18: Serotype 14: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 14 | 73.9639 (29.28795)
  21-day dosing schedule: Week 18: Serotype 17: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 17 | 76.0492 (42.17688)
  21-day dosing schedule: Week 18: Serotype 19: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 19 | 94.4390 (30.99072)
  21-day dosing schedule: Week 18: Serotype 2: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 2 | 80.1377 (36.22955)
  21-day dosing schedule: Week 18: Serotype 20: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 20 | 83.5202 (42.23144)
  21-day dosing schedule: Week 18: Serotype 22: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 22 | 91.9216 (20.16314)
  21-day dosing schedule: Week 18: Serotype 23: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 23 | 84.5653 (31.15550)
  21-day dosing schedule: Week 18: Serotype 26: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 26 | 88.7836 (30.46916)
  21-day dosing schedule: Week 18: Serotype 3: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 3 | 90.4017 (39.81294)
  21-day dosing schedule: Week 18: Serotype 34: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 34 | 91.6269 (16.96157)
  21-day dosing schedule: Week 18: Serotype 4: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 4 | 79.5022 (41.16158)
  21-day dosing schedule: Week 18: Serotype 43: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 43 | 81.6962 (28.91186)
  21-day dosing schedule: Week 18: Serotype 5: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 5 | 88.6356 (17.56577)
  21-day dosing schedule: Week 18: Serotype 51: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 51 | 71.0749 (31.74626)
  21-day dosing schedule: Week 18: Serotype 54: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 54 | 72.7200 (31.26330)
  21-day dosing schedule: Week 18: Serotype 56: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 56 | 82.4508 (27.11113)
  21-day dosing schedule: Week 18: Serotype 57: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 57 | 98.1611 (9.69314)
  21-day dosing schedule: Week 18: Serotype 68: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 68 | 82.9015 (37.95746)
  21-day dosing schedule: Week 18: Serotype 70: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 70 | 91.3286 (19.12896)
  21-day dosing schedule: Week 18: Serotype 8: number analyzed (Participants) | 3
  21-day dosing schedule: Week 18: Serotype 8 | 65.5637 (36.02827)
  21-day dosing schedule: Week 18: Serotype 9: number analyzed (Participants) | 4
  21-day dosing schedule: Week 18: Serotype 9 | 75.8333 (30.77330)

ADVERSE EVENTS:
Time Frame: Up to study termination visit (Week 52)
Description: The SAF included all participants who had received at least 1 dose of study medication.
Arm/Group | Kedrion IVIG 10%
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 4/47
Other Adverse Events (participants affected / at risk) | 38/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kedrion IVIG 10% (N=47)
Cholecystitis acute (Hepatobiliary disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kedrion IVIG 10% (N=47)
Headache (Nervous system disorders) | 19
Fatigue (General disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Sinusitis (Nervous system disorders) | 11
upper respiratory tract infection (Infections and infestations) | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 6
Coombs direct test positive (Investigations) | 6
Depression (Psychiatric disorders) | 6
Bronchitis (Infections and infestations) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Influenzae (Infections and infestations) | 3
Dizziness (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Chills (General disorders) | 3
Pain (General disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Skin laceration (Injury, poisoning and procedural complications) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Insomnia (Psychiatric disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Investigators can be divulged to third parties from the trial team only after Kedrion's approval.

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03961009/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT03961009/SAP_001.pdf